CLINICAL TRIAL: NCT03952624
Title: Patient-Centered Assessment of Symptoms and Outcomes
Status: Recruiting | Type: Observational
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 190098; 19-NR-0098
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12-22

CONDITIONS: Fatigue; Cancer; CFS; ME/CFS; Myalgic Encephalomyelitis/Chronic Fatigue Syndrome; Lupus; Systemic Lupus Erthematosus; Sjogrens
Keywords: Symptom Biology; Symptom Phenotyping; Fatigue; Natural History
MeSH Terms: conditions — Fatigue; Neoplasms; Fatigue Syndrome, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: FNS <= 3
- Fatigued: FNS >= 4

SUMMARY:
Background:

The cause of fatigue is not well understood. It can be felt differently by different people. Some people think there are different types of fatigue, with different causes. Researchers think a therapy to treat one type of fatigue in one condition should be able to treat that type of fatigue in other conditions.

Objective:

To understand the types of fatigue.

Eligibility:

Adults 18 and older who have felt fatigue for more than a month, and non-fatigued adults

Design:

Participants will be screened with a physical exam, their medical history, a vision test, and blood and urine tests.

Participants will begin to track the foods they eat.

This study will involve up to 10 visits. Each visit will last no more than 4 hours.

In Stage 1, participants will have an interview, fill out questionnaires, and play computer games. They will take walking and handgrip tests. They will give blood, urine, and saliva samples. They will wear a wrist monitor at home for 7 days and write down their activities. They will be put into a group: fatigue or non-fatigued control.

In Stage 2, participants will answer questionnaires and give a blood sample. They will have heart tests. They may take exercise and lung function tests that include wearing a nose clip. They may have an optional brain MRI: They may wear an electrode cap on their head during the scan to measure brain activity. They will lie on table that slides into a cylinder. They may perform tasks in the scanner.

After the study, participants might be contacted about other studies.

...

DETAILED DESCRIPTION:
Purpose: The purpose of this study is to allow for deep and broad phenotyping of persons with clinically-meaningful fatiguing symptoms, regardless of physiologic or pathologic condition. This protocol will enable the National Institute of Nursing Research (NINR) investigators to describe the clinical characteristics of persons reporting clinically-meaningful fatigue and collect clinical and scientific data for the purpose of making comprehensive phenotypic descriptions.

These phenotypic descriptions will be used to explore the heterogeneity of fatiguing symptoms to clarify the nature of different fatigue phenotypes and their biologic correlates.

The specific goals of this protocol are the following:

* To characterize and phenotype individuals with clinically-meaningful fatigue.
* To explore the heterogeneity of fatiguing conditions to define specific fatigue dimensions.
* To generate hypotheses of the possible mechanism of each fatigue dimension.

Study Population: The study population will consist of up to 692 persons with or without clinically-meaningful fatigue. Approximately 20 will be enrolled in the technical development sub-study to refine the neuroimaging techniques used in this study. Additional 20 healthy volunteers will be enrolled to serve as normative reference. This protocol is open to anyone of any ethnicity, sex, or nationality.

Design: The protocol is designed as an exploratory multi-stage study. Upon receiving inquiry from a potential participant, a phone screening using an eligibility questionnaire and an in-person NIH outpatient screening visit will be conducted. If a treatable medical condition is identified during the screening that directly contributes to the fatigue experience, then the participant will not proceed in the study but will be asked to see their care provider for evaluation and/or management. Those who are under a known treatment (e.g., chemotherapy, antivirals) for a clinical condition or those without a clear clinical explanation for their fatigue will be invited to participate in Stage 1 of the study. Stage 1 is the fatigue assessment stage and includes completion of self-report questionnaires and performance tasks. Stage 2 will include additional clinical and scientific assessments to allow for deeper understanding of the fatigue phenotype.

Before study termination, participants may be referred to appropriate NIH CC services for management recommendations. Participants who complete the study may be re-contacted about other available fatigue intervention studies.

Multi-Stage Study Design

Stage 1 - Fatigue Assessment

Stage 2 - Fatigue Dimension Phenotyping Evaluation

Outcome Measures: The study will use a wide variety of measurement tools for phenotyping purposes. These include: vital signs, medical history, physical exam, blood draw, medical record review, clinical interviews, patient reported outcome measurements, physical, cognitive, affective, and behavioral measurements, structural and functional imaging assessments, nutritional assessment, clinical and research laboratory measurements, and electrocardiogram.

In summary, the NINR Patient-Centered Assessment of Symptoms and Outcomes (P-CASO) protocol will enable investigators to obtain detailed clinical descriptions and to collect phenotyping measurements from research participants who report clinically-meaningful fatigue.

The study will allow NINR investigators to perform descriptive research on fatigue for hypothesis generation.

ELIGIBILITY:
* INCLUSION CRITERIA:

All Participants (including returning participants)

* Adult participants aged >= 18 years at the time of enrollment.
* Able to provide written informed consent.
* Willing and able to complete study procedures.

Fatigued Participants

-In addition to the above, must experience fatigue for more than a month.

Healthy Volunteers for the fMRI study

* Right handed
* Not taking any prescribed medications for chronic medical conditions
* Not diagnosed with any chronic medical condition

EXCLUSION CRITERIA:

Exclusion from study entry:

* Not fluent in English.
* Have medical health issues that create additional and substantial adverse risks related to study procedures. Medical examples are the acute complications of medical disease, such as unstable hypertension, diabetic ketoacidosis, symptomatic hyperthyroidism, and unstable angina.
* Have a psychiatric condition that prevents participant from being able to reliably report the fatigue experience (e.g., a psychotic disorder with severely disorganized thinking);
* Current substance use disorder within the last five years or positive urine toxicology results at enrollment and before Stage 2. Prior marijuana use within the past five years will not be an exclusion.
* Categorized as a high-risk drinker (>=5 drinks/day and >=15 drinks/week for men, >=4 drinks/day and >=8 drinks/week for women). ( Dietary Guidelines for Americans 2015-2020," U.S. Department of Health and Human Services and U.S. Department of Agriculture).
* NIH employees.
* Pregnant or lactating women.
* Ongoing medical condition that is deemed by the Principal Investigator to interfere with the conduct or assessments of the study or safety of the participant.

Exclusion from specific tests:

* fMRI Technical Development Sub-Study

  * Implanted cardiac pacemakers, metal aneurysm clips;
  * Broken bones repaired with metal pins, screws, rods, plates;
  * Prosthetic eye implants;
  * Transdermal medications or infusion pumps;
  * Bullet fragments or other metal pieces in body from old wounds;
  * Significant work exposure to metal particles;
  * Clinically relevant claustrophobia;
  * Unable to lie comfortably on back for up to 4 hours;
  * Left-handed. (Participants that are ambidextrous, will complete the Edinburgh Handedness Inventory).
* EEfRT and Stroop Test

  * Severe essential hand tremor or severe hand pain (e.g., severe arthritis or severe carpel tunnel) that makes it difficult to perform rapid keyboard presses will be an exclusion from the EEfRT and Stroop Test.
  * Color-blindness, verified by scoring >14 on the Ishihara card test, will exclude a participant from taking the Stroop test. The Ishihara card test will be administered only if the participant states he or she is color-blind.
* Tilt Table Test

  --Beta blocker medications.
* CPET

  * Any neuromuscular conditions (e.g., multiple sclerosis, Parkinson s disease) with significant mobility impairment that prohibits treadmill or bike performance, or any medical condition (e.g., congestive heart failure, coronary artery disease, chronic obstructive pulmonary disease [COPD], severe osteoarthritis and poorly controlled asthma) that would make it risky for the participant to exercise (e.g., exercise-induced angina and asthma), will exclude a participant from the CPET.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited via a stepwise approach. Limited recruitment will occur during the first 6 months to 12 months after initial IRB approval, as part of the feasibility assessment. During this time, NIH investigators such as those from NINR, the NIDCR Sjogren s Clinic, and the 16-N-0058 study (Myalgic Encephalomyelitis/Chronic Fatigue Syndrome) will be informed about the study. These investigators will not actively recruit their own patients for the study but will be asked to post a recruitment flyer in their clinics. After the first year, the study will open to the general population.
Sampling Method: Non-Probability Sample
Enrollment: 692 (Estimated)
Dates: Start 2019-09-13 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Fatigue Level | Stage 1 and Stage 2
  The primary outcome will be the fatigue level using the Fatigue Numeric Rating Scale (FNS) score.

SECONDARY OUTCOMES:
Secondary outcomes of the study will obtain common fatigue dimension information from participants that will allow us to better define phenotypic clusters that ultimately can be used for hypothesis generation, these include patient-reported outc... | All time points

CONTACTS AND LOCATIONS:
Overall Officials: Miroslav Backonja, M.D., Principal Investigator — National Center for Complementary and Integrative Health (NCCIH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Saligan LN, Olson K, Filler K, Larkin D, Cramp F, Yennurajalingam S, Escalante CP, del Giglio A, Kober KM, Kamath J, Palesh O, Mustian K; Multinational Association of Supportive Care in Cancer Fatigue Study Group-Biomarker Working Group. The biology of cancer-related fatigue: a review of the literature. Support Care Cancer. 2015 Aug;23(8):2461-78. doi: 10.1007/s00520-015-2763-0. Epub 2015 May 15. PMID 25975676
- [Background] Ramsey-Goldman R, Rothrock N. Fatigue in systemic lupus erythematosus and rheumatoid arthritis. PM R. 2010 May;2(5):384-92. doi: 10.1016/j.pmrj.2010.03.026. PMID 20656619
- [Background] Sharpe M, Wilks D. Fatigue. BMJ. 2002 Aug 31;325(7362):480-3. doi: 10.1136/bmj.325.7362.480. No abstract available. PMID 12202331
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2019-NR-0098.html